CLINICAL TRIAL: NCT00476060
Title: Autologous Mesenchymal Stem Cell Transplantation in Patients With Decompensated Cirrhosis: A Randomized Placebo-controlled Trial
Brief Title: Mesenchymal Stem Cell Transplantation in Decompensated Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Tehran (Other)
Responsible Party: Principal Investigator, Mehdi Mohamadnejad, Assistant Professor of Medicine, University of Tehran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DDRC85-13
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Cirrhosis
Keywords: Cirrhosis; Bone marrow; Mesenchymal stem cell; MELD score; Quality of life
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Procedure: Autologous mesenchymal stem cell transplantation
- B (Placebo Comparator)
  Interventions: Procedure: Autologous mesenchymal stem cell transplantation

INTERVENTIONS:
Procedure: Autologous mesenchymal stem cell transplantation — Arm A: 300 million cells will be infused one time through a peripheral vein/// Arm B: Infusion of placebo one time through a peripheral vein

SUMMARY:
The standard treatment for decompensated cirrhosis is liver transplantation, however, it has several limitations. Recent animal studies suggest that bone marrow stem cell transplantation can lead to regression of liver fibrosis. The investigators have already completed the phase 1 study of bone marrow mesenchymal stem cell (MSC) transplantation in 4 patients with cirrhosis. The procedure was safe, and feasible, and led to somewhat promising results (Mohamadnejad M, et al. 2006; Submitted for publication). The aim of this study is to find efficacy of this new treatment strategy in the setting of a multicenter, randomized placebo-controlled trial in 50 patients with decompensated cirrhosis.

DETAILED DESCRIPTION:
The standard treatment for decompensated cirrhosis is liver transplantation, however, it has several limitations, including small donor pool, long waiting list, and several complications. Recent animal studies suggest that bone marrow stem cell transplantation can lead to regression of liver fibrosis. The investigators have already completed the phase 1 study of bone marrow mesenchymal stem cell (MSC) transplantation in 4 patients with cirrhosis. The procedure was safe, and feasible, and led to somewhat promising results (Mohamadnejad M, et al. 2006; Submitted for publication). The aim of this study is to find efficacy of this new treatment strategy in the setting of a multicenter, randomized placebo controlled trial. After assignment of the written informed consent, thirty six patients with decompensated cirrhosis will be enrolled, and will be randomized by block randomization into treatment or placebo arm. All the enrolled patients will be in the waiting list of liver transplantation. In the treatment arm bone marrow of the patients will be aspirated, and autologous bone marrow mesenchymal stem cells will be cultured, and then will be infused through a peripheral vein. Also, the corresponding placebo will be infused for the placebo group. The patients will be followed up for 1 year after performing the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis (diagnosed by clinical, biochemical, sonographic, and histologic evidences of cirrhosis) (Patients will have histological documentation of cirrhosis before enrollment. However, for those with evidences of severe coagulopathy liver biopsy may not be performed)
* Evidences of decompensated liver disease at screening (e.g. child class B, or C)

Exclusion Criteria:

* Presence of active hepatic encephalopathy
* Refractory ascites
* Evidences of active autoimmune liver disease (e.g. gamma globulin of more than 2 times of upper limit of normal, and ALT > 3 times normal in patients with autoimmune hepatitis)
* Hepatocellular carcinoma or other malignancies
* Active infectious disease
* Presences of severe underlying cardiac, pulmonary, or renal disease
* Alcohol use in the last 3 months before screening
* Use of hepatotoxic drugs in the last 3 months before screening
* Unwilling to assign the informed consent
* Presence of significant extrahepatic biliary disease (e.g. CBD stone, PSC, etc.)
* Positive HIV ab
* Positive HBsAg with detectable HBV DNA PCR
* Positive HCV Ab with detectable HCV RNA PCR
* Active thrombosis of the portal or hepatic veins
* Serum Cr > 1.8 mg/dL at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
MELD score, quality of life, liver volume, histological improvement (In a subset of patients with evidences of clinical and biochemical improvement, follow up liver biopsy will be performed at the end of follow up). | One year

SECONDARY OUTCOMES:
All cause mortality, tracking the infused cells in the patients' bodies. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Reza Malekzadeh, M.D, Study Chair — Digestive Disease Research Center, Medical Sciences/ University of Tehran; Ardeshir Ghavamzadeh, M.D., Study Chair — Hematology, Oncology, and BMT research center, Medical Sciences/University of Tehran; Mehdi Mohamadnejad, M.D., Principal Investigator — Digestive Disease Research Center, Medical Scineces/ University of Tehran; Kamran Alimoghaddam, M.D., Principal Investigator — Hematology, Oncology, and BMT research center, Medical Sciences/University of Tehran
Locations (1):
- Digestive Disease Research Center, Shariati Hospital, Tehran, Iran